CLINICAL TRIAL: NCT04544904
Title: Novel Uses of Technology for Individuals With Mild to Moderate Hip or Knee Osteoarthritis: The Technology, Exercise Programming, and Activity Prescription for Enhanced Mobility (TEAM) Study
Brief Title: The Technology, Exercise Programming, and Activity Prescription for Enhanced Mobility (TEAM) Study
Acronym: TEAM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020TEAM
Record Dates: First submitted 2020-08-24; First posted 2020-09-10 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Osteo Arthritis Knee; Osteoarthritis; Hip Arthritis
Keywords: exercise; physical activity; medicine
MeSH Terms: conditions — Osteoarthritis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Patients will receive the usual care.
- PAARx (Experimental): Patients will be prescribed technology-based physical activity programming.
  Interventions: Device: PAARx
- PAARx and JM (Experimental): Patients will be prescribed technology-based physical activity programming and be referred to a web-based resource for evidence-based joint management.
  Interventions: Device: PAARx; Device: JM

INTERVENTIONS:
Device: PAARx — Prescription Physical Activity Programming Application
  Arms: PAARx; PAARx and JM
Device: JM — Joint Management (JM) web-based joint management resource.
  Arms: PAARx and JM

SUMMARY:
Many individuals with osteoarthritis (OA) (up to 45%) are referred to an orthopaedic surgeon for a joint replacement prematurely or will not be candidates for surgery. These individuals need appropriate (non-operative) care to help reduce their pain and enhance their mobility. We are studying the use of innovative technology to help physicians give physical activity advice for patients to become more active and provide free online resources to help patients understand OA self-management and exercise, especially when they have barriers to accessing formal care. Individuals with OA that are referred to a specialized clinic will receive one of three interventions: usual care (handout on resources), a physical activity prescription by a doctor, or the prescription and a link to a free web-based platform (website) on non-operative management of OA with patient education and exercise videos. Our goal is to help with non-operative management strategies to improve quality of life, reduce pain, improve mobility, and possibly delay or prevent a joint replacement.

Osteoarthritis is a condition where people feel joint pain or stiffness. Joints are the body parts where two bones join together with softer material (cartilage) between them. In osteoarthritis, this cartilage wears down. It is the biggest cause for disability worldwide. Helping people with osteoarthritis starts with education, physical activity, and physiotherapy. Doctors can also prescribe braces, injections or medications. For severe osteoarthritis when nothing else helps, surgery can be done to replace the joint.

Doctors often refer patients for surgery too soon. Skipping steps of care may mean unnecessary surgery and longer wait times. The Musculoskeletal Rapid Access Clinic (now called Clinic) in London was set up to solve these problems. They screen patients before referring them to a surgeon, and do not refer almost half of patients. Our goal is to support these patients with new ways to make their non-surgical treatment better.

The first way is through physical activity 'prescription'. It works well for other chronic conditions and patients say it helps. We don't know how well it works for people with osteoarthritis. Most doctors have little time, training or experience for prescribing physical activity. Technology can make it easier for doctors and patients. We have designed a tool to help doctors prescribe physical activity and a smartphone app to track patient activity. We have also created a free website. This includes patient education, exercise videos, and virtual physiotherapy. This can be important for individuals who can't access in-person care.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the leading cause of disability worldwide and affects more than 4.4 million Canadians. Current evidence-based guidelines for OA management recommend weight management, patient education, physical activity, physiotherapy (PT), bracing, viscosupplementation, and anti-inflammatory/pain medications prior to joint replacement surgery. Unfortunately, current practice trends are not consistent with these guidelines, as nearly half of patients with OA referred to orthopedic surgeons do not require total joint arthroplasty (TJA) at the time of initial consultation. Through the Southwest Musculoskeletal Rapid Access Clinic (RAC), approximately ten referrals (20%) are rejected each day due to OA criteria not met, and a further 20% are assessed as non-operative.

We aim to identify individuals with 'mild to moderate' OA and optimize their first-line non-operative management, starting with physical activity and education.

Physical activity prescriptions are effective in increasing patient levels of physical activity, and 93% of patients surveyed want advice on physical activity from their physicians; but it is underused.

Physicians cite lack of time and inadequate training as barriers. Electronic screening of physical activity behaviours can save time for physicians, and the use of digital health tools can improve physical activity levels.

Patient education and physiotherapist-led group exercise therapy programs have shown to delay progression of knee OA symptoms and improve pain and function; however, two of the most significant barriers to accessing exercise programming is the cost (~approximate $425-475 per 6-8-week session) and accessibility to attend the exercise session (proximity to facility, remote/rural communities, etc.).

The Need for a Solution that targets both Providers and Patients Screening for baseline physical activity levels and including educational components significantly increase intervention effectiveness.

We have previously tested the feasibility of implementing an e-health tool to support physical activity counselling by physicians during patients' periodic health review. We will adapt and implement this tool, Physical Activity and App Prescription (PARx) to screen and provide tailored resources for physical activity in the setting of OA. We will use tablet computers and email, directly linked with the electronic medical record (EMR), to engage patients in contemplating their own physical activity levels, start conversations with their healthcare providers (in this case, primary care physicians with additional training in sport and exercise medicine), and support customized, patient-centered health care. After patients enter their information, they will receive evidence-based behavioural change supports to help them meet their goals.

The automated algorithm assesses current activity level, risk factors/comorbidities and readiness for change. Based on the answers provided, patients are risk-stratified and tailored resources will be provided to the patient and to their clinician in the form of decision support tools embedded in the EMR. This will include the novel implementation of an exercise tracking platform via the smartphone app (myrecovery.ai).

The web-based platform Joint Management (JM) is a free, readily accessible evidenced-based resource focusing on non-operative management strategies for mild to moderate hip and knee OA. The platform will include exercise programming (videos, pictures, and descriptions of the exercises) and patient education (benefits of exercise, lifestyle modifications, nutrition, injections, etc.), to assist the patient engage in self-management. JM will also include the option for (paid) virtual access to PTs, who can provide individualized support, recommendations and exercise programming via the platform.

RATIONALE:

Creating customized physical activity plans with automated reminders and other supports addresses the problem of self-efficacy in providers by developing an evidence-based automated method, while also addressing the issue of patient adherence by using tailored behaviour change techniques, through assessing readiness for change, and helping patients create new habits.

The motivation for JM is to create a free, online evidence-based OA education and exercise programming resource for those that are not able to afford or access community-based exercise programs. The virtual PT option will help optimize patient's experience with the web-based platform, offering support and personalized recommendations regarding management of their condition and exercise programming tailored to their specific abilities, preferences, and needs.

Why this is Innovative:

The evidence for using patient-reported measures and functional outcomes to guide quality improvement for personalized OA care in a systematic manner is in an early stage, meaning that this project can not only impact healthcare delivery and translate new knowledge into medical practice but help position Western University as a leader in this area. The novel technologies (PARx and JM) are innovative tools informed by patient priorities and co-designed with our patient partners, specifically geared towards 1) developing new and more personalized treatment approaches, 2) developing more effective self-management tools, and 3) reducing disparities in vulnerable and hard-to-reach populations. To this end, we will share our findings broadly with our patient partners and reach out to these harder-to-reach groups in particular.

EXPECTED OUTCOMES:

Health Outcomes: We expect to increase patients' physical activity and improve outcomes for individuals with mild to moderate OA. We aim to optimize non-operative management of OA symptoms and therefore possibly delay and/or prevent the need for TJA.

Academic Outcomes: We expect to develop a model of physical activity prescription and patient education that can be scaled up for implementation in primary care.

Societal Outcomes: Both novel technologies have the potential to be implemented across Canada, targeting modifying disease progression and, ideally, delaying or preventing TJA.

Innovative Technology 1: Physical Activity (PA) and App Prescription (Rx) (PARx) Physical Activity and App Prescription (PARx): Tablet/email software (REDCap) is used to collect physical activity data from patient input and prompt intervention by providers. The automated algorithm assesses current activity level, risk factors/comorbidities and readiness for change. Based upon their answers, patients will be risk-stratified and tailored resources will be provided to them in the form of a personalized prescription and free smartphone app (myrecovery.ai) to track activity levels.

Innovative Technology 2: Joint Management (JM) Joint Management (JM): This is a free online evidence-based OA education and exercise programming resource for those that are not able to afford or access community-based exercise programs, with a virtual physiotherapy (PT) option to offer support and personalized recommendations.

OBJECTIVES:

The objective of the proposed study is to 1) determine if PARx and JM will improve pain, increase physical activity levels, and improve functional outcomes in patients with mild to moderate hip or knee OA

RESEARCH QUESTIONS:

1. Does the use of novel technology (PARx) affect patient reported outcomes in individuals with mild to moderate hip or knee OA?
2. Does PARx influence activity levels in individuals with mild to moderate hip or knee OA?
3. Does the use of novel technology (PARx and JM) affect patient reported and functional outcomes in individuals with mild to moderate hip or knee OA?
4. What are the experiences and perceptions of patients and physicians during this process?

SPECIFIC AIMS:

Measure and compare A1) patient reported outcomes (pain, joint stiffness, disability, quality of life, disease knowledge, self-efficacy, depression, and fatigue), A2) physical activity levels, and A3) functional outcomes with those that have access (PARx and JM) and those that do not have access (usual care) to the technology. Determine A4) participant and physician experiences.

HYPOTHESES:

We hypothesize that access to technology-facilitated physical activity prescription (PARx) and access to the web-based platform (JM) will H1) improve patient reported outcomes (pain, joint stiffness, disability, quality of life, disease knowledge, self-efficacy, depression, and fatigue), H2) increase PA levels, and H3) improve functional outcomes in individuals with mild to moderate hip or knee OA compared to usual care. We hypothesize that access to JM will result in a greater improvement than PARx alone.

ELIGIBILITY:
Inclusion Criteria:

* 40-74 years of age
* Screened by the Southwest Musculoskeletal RAC as "mild to moderate OA" using clinical and radiographic criteria

Exclusion Criteria:

* Concomitant end-stage OA (awaiting/prior TJA)
* Inflammatory arthritis (rheumatoid, psoriatic, or disease-modifying anti-rheumatic drug exposure)
* Unstable medical conditions that would preclude physical activity prescription (e.g. unstable angina, uncontrolled Type 2 Diabetes)
* Not able/willing to follow up for the study period
* Does not have access to the internet
* Cannot communicate in English.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2025-06-06 (Estimated); Study Completion 2025-06-06 (Estimated)

PRIMARY OUTCOMES:
height | Baseline
  height in cm
height | 2 months
  height in cm
height | 6 months
  height in cm
height | 12 months
  height in cm
body mass index (derived) | Baseline
  body mass index as calculated with height and weight
body mass index (derived) | 2 months
  body mass index as calculated with height and weight
body mass index (derived) | 6 months
  body mass index as calculated with height and weight
body mass index (derived) | 12 months
  body mass index as calculated with height and weight
abdominal circumference | Baseline
  abdominal circumference in cm
abdominal circumference | 2 months
  abdominal circumference in cm
abdominal circumference | 6 months
  abdominal circumference in cm
abdominal circumference | 12 months
  abdominal circumference in cm
weight | Baseline
  weight kg
  , weight, body mass index (derived), abdominal circumference, and medical history to assess for comorbid disease.
weight | 2 months
  weight kg
  , weight, body mass index (derived), abdominal circumference, and medical history to assess for comorbid disease.
weight | 6 months
  weight kg
  , weight, body mass index (derived), abdominal circumference, and medical history to assess for comorbid disease.
weight | 12 months
  weight kg
  , weight, body mass index (derived), abdominal circumference, and medical history to assess for comorbid disease.
PA Evaluation | Baseline
  PA levels will be measured as a composite measure using smartphone app/accelerometer data (myrecovery.ai; steps per day, light/moderate/vigorous activity, and total MET-min) via the International PA Questionnaire - Short Form (IPAQ-SF) [15].
PA Evaluation | 2 months
  PA levels will be measured as a composite measure using smartphone app/accelerometer data (myrecovery.ai; steps per day, light/moderate/vigorous activity, and total MET-min) via the International PA Questionnaire - Short Form (IPAQ-SF) [15].
PA Evaluation | 6 months
  PA levels will be measured as a composite measure using smartphone app/accelerometer data (myrecovery.ai; steps per day, light/moderate/vigorous activity, and total MET-min) via the International PA Questionnaire - Short Form (IPAQ-SF) [15].
PA Evaluation | 12 months
  PA levels will be measured as a composite measure using smartphone app/accelerometer data (myrecovery.ai; steps per day, light/moderate/vigorous activity, and total MET-min) via the International PA Questionnaire - Short Form (IPAQ-SF) [15].
Functional Assessment 30 second sit-to-stand test | Baseline
  30 second sit-to-stand test
Functional Assessment 30 second sit-to-stand test | 2 months
  30 second sit-to-stand test
Functional Assessment 30 second sit-to-stand test | 6 months
  30 second sit-to-stand test
Functional Assessment 30 second sit-to-stand test | 12 months
  30 second sit-to-stand test
Functional Assessment 40-meter fast-paced walk test | Baseline
  40-meter fast-paced walk test
Functional Assessment 40-meter fast-paced walk test | 2 months
  40-meter fast-paced walk test
Functional Assessment 40-meter fast-paced walk test | 6 months
  40-meter fast-paced walk test
Functional Assessment 40-meter fast-paced walk test | 12 months
  40-meter fast-paced walk test
Hip Disability and OA Outcome Score (HOOS) | Baseline
  Hip Disability and Osteoarthritis Outcome Score (HOOS) assesses patient pain (10 items), satisfaction including stiffness and range of motion (5 items), activity limitations-daily living (17 items), sports and recreation function (4 items), and hip related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible hip symptoms and 100 indicating no hip symptoms. This is a patient reported joint-specific score, which may be useful for assessing changes in hip pathology over time, with or without treatment.
Hip Disability and OA Outcome Score (HOOS) | 2 months
  Hip Disability and Osteoarthritis Outcome Score (HOOS) assesses patient pain (10 items), satisfaction including stiffness and range of motion (5 items), activity limitations-daily living (17 items), sports and recreation function (4 items), and hip related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible hip symptoms and 100 indicating no hip symptoms. This is a patient reported joint-specific score, which may be useful for assessing changes in hip pathology over time, with or without treatment.
Hip Disability and OA Outcome Score (HOOS) | 6 months
  Hip Disability and Osteoarthritis Outcome Score (HOOS) assesses patient pain (10 items), satisfaction including stiffness and range of motion (5 items), activity limitations-daily living (17 items), sports and recreation function (4 items), and hip related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible hip symptoms and 100 indicating no hip symptoms. This is a patient reported joint-specific score, which may be useful for assessing changes in hip pathology over time, with or without treatment.
Hip Disability and OA Outcome Score (HOOS) | 12 months
  Hip Disability and Osteoarthritis Outcome Score (HOOS) assesses patient pain (10 items), satisfaction including stiffness and range of motion (5 items), activity limitations-daily living (17 items), sports and recreation function (4 items), and hip related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible hip symptoms and 100 indicating no hip symptoms. This is a patient reported joint-specific score, which may be useful for assessing changes in hip pathology over time, with or without treatment.
Knee OA Outcome Score (KOOS) | Baseline
  Knee injury and Osteoarthritis Outcome Score (KOOS) assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms. The KOOS is a patient reported joint-specific score, which may be useful for assessing changes in knee pathology over time, with or without treatment.
Knee OA Outcome Score (KOOS) | 2 months
  Knee injury and Osteoarthritis Outcome Score (KOOS) assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms. The KOOS is a patient reported joint-specific score, which may be useful for assessing changes in knee pathology over time, with or without treatment.
Knee OA Outcome Score (KOOS) | 6 months
  Knee injury and Osteoarthritis Outcome Score (KOOS) assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms. The KOOS is a patient reported joint-specific score, which may be useful for assessing changes in knee pathology over time, with or without treatment.
Knee OA Outcome Score (KOOS) | 12 months
  Knee injury and Osteoarthritis Outcome Score (KOOS) assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms. The KOOS is a patient reported joint-specific score, which may be useful for assessing changes in knee pathology over time, with or without treatment.
Intermittent and Constant OA Pain (ICOAP) | Baseline
  This 11-item tool is designed to assess pain in individuals with hip or knee osteoarthritis taking into account both constant and intermittent pain experiences. There are two versions of this tool; one to assess pain in the knee joint and another assessing pain in the hip joint.
Intermittent and Constant OA Pain (ICOAP) | 2 months
  This 11-item tool is designed to assess pain in individuals with hip or knee osteoarthritis taking into account both constant and intermittent pain experiences. There are two versions of this tool; one to assess pain in the knee joint and another assessing pain in the hip joint.
Intermittent and Constant OA Pain (ICOAP) | 6 months
  This 11-item tool is designed to assess pain in individuals with hip or knee osteoarthritis taking into account both constant and intermittent pain experiences. There are two versions of this tool; one to assess pain in the knee joint and another assessing pain in the hip joint.
Intermittent and Constant OA Pain (ICOAP) | 12 months
  This 11-item tool is designed to assess pain in individuals with hip or knee osteoarthritis taking into account both constant and intermittent pain experiences. There are two versions of this tool; one to assess pain in the knee joint and another assessing pain in the hip joint.
Patient Global Assessment of Health Status (PGA) | Baseline
  Patient global assessment (PGA) is one of the most widely used PROs in RA practice and research and is included in several composite scores such as the 28-joint Disease Activity Score (DAS28). PGA is often assessed by a single question with a 0-10 or 0-100 response.
Patient Global Assessment of Health Status (PGA) | 2 months
  Patient global assessment (PGA) is one of the most widely used PROs in RA practice and research and is included in several composite scores such as the 28-joint Disease Activity Score (DAS28). PGA is often assessed by a single question with a 0-10 or 0-100 response.
Patient Global Assessment of Health Status (PGA) | 6 months
  Patient global assessment (PGA) is one of the most widely used PROs in RA practice and research and is included in several composite scores such as the 28-joint Disease Activity Score (DAS28). PGA is often assessed by a single question with a 0-10 or 0-100 response.
Patient Global Assessment of Health Status (PGA) | 12 months
  Patient global assessment (PGA) is one of the most widely used PROs in RA practice and research and is included in several composite scores such as the 28-joint Disease Activity Score (DAS28). PGA is often assessed by a single question with a 0-10 or 0-100 response.
Patient Acceptable Symptom State (PASS) | Baseline
  Patient Acceptable Symptom State (PASS) has been defined as the highest level of symptom beyond which patients consider themselves well.
Patient Acceptable Symptom State (PASS) | 2 months
  Patient Acceptable Symptom State (PASS) has been defined as the highest level of symptom beyond which patients consider themselves well.
Patient Acceptable Symptom State (PASS) | 6 months
  Patient Acceptable Symptom State (PASS) has been defined as the highest level of symptom beyond which patients consider themselves well.
Patient Acceptable Symptom State (PASS) | 12 months
  Patient Acceptable Symptom State (PASS) has been defined as the highest level of symptom beyond which patients consider themselves well.
Arthritis Self-Efficacy Questionnaire | Baseline
  The ASES was developed to measure patients' arthritis-specific self-efficacy, or patients' beliefs that they could perform specific tasks or behaviors to cope with the consequences of arthritis.
Arthritis Self-Efficacy Questionnaire | 2 months
  The ASES was developed to measure patients' arthritis-specific self-efficacy, or patients' beliefs that they could perform specific tasks or behaviors to cope with the consequences of arthritis.
Arthritis Self-Efficacy Questionnaire | 6 months
  The ASES was developed to measure patients' arthritis-specific self-efficacy, or patients' beliefs that they could perform specific tasks or behaviors to cope with the consequences of arthritis.
Arthritis Self-Efficacy Questionnaire | 12 months
  The ASES was developed to measure patients' arthritis-specific self-efficacy, or patients' beliefs that they could perform specific tasks or behaviors to cope with the consequences of arthritis.
Center for the Epidemiological studies - Depression Scale (CES-D) | Baseline
  The Center for Epidemiologic Studies Depression Scale is a commonly used freely available self-report measure of depressive symptoms.
Center for the Epidemiological studies - Depression Scale (CES-D) | 2 months
  The Center for Epidemiologic Studies Depression Scale is a commonly used freely available self-report measure of depressive symptoms.
Center for the Epidemiological studies - Depression Scale (CES-D) | 6 months
  The Center for Epidemiologic Studies Depression Scale is a commonly used freely available self-report measure of depressive symptoms.
Center for the Epidemiological studies - Depression Scale (CES-D) | 12 months
  The Center for Epidemiologic Studies Depression Scale is a commonly used freely available self-report measure of depressive symptoms.
Visual Analogue Scale to Evaluate Fatigue Severity (VAS-F) | Baseline
  The scale consists of 18 items relating to the subjective experience of fatigue. Each item asks respondents to place an "X," representing how they currently feel, along a visual analogue line that extends between two extremes (e.g., from "not at all tired" to "extremely tired").
Visual Analogue Scale to Evaluate Fatigue Severity (VAS-F) | 2 months
  The scale consists of 18 items relating to the subjective experience of fatigue. Each item asks respondents to place an "X," representing how they currently feel, along a visual analogue line that extends between two extremes (e.g., from "not at all tired" to "extremely tired").
Visual Analogue Scale to Evaluate Fatigue Severity (VAS-F) | 6 months
  The scale consists of 18 items relating to the subjective experience of fatigue. Each item asks respondents to place an "X," representing how they currently feel, along a visual analogue line that extends between two extremes (e.g., from "not at all tired" to "extremely tired").
Visual Analogue Scale to Evaluate Fatigue Severity (VAS-F) | 12 months
  The scale consists of 18 items relating to the subjective experience of fatigue. Each item asks respondents to place an "X," representing how they currently feel, along a visual analogue line that extends between two extremes (e.g., from "not at all tired" to "extremely tired").

CONTACTS AND LOCATIONS:
Overall Officials: Jane Thornton, MD PhD, Principal Investigator — Western University
Locations (1):
- Fowler Kennedy Sports Medicine Clinic, London, Ontario, Canada

REFERENCES:
- [Background] Bombardier, C., G. Hawker, and D. Mosher, The Impact of Arthritis in Canada: Today and Over the Next 30 Years. 2011, Arthritis Alliance of Canada: Canadian Arthritis Network.
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] King LK, Marshall DA, Faris P, Woodhouse LJ, Jones CA, Noseworthy T, Bohm E, Dunbar MJ, Hawker GA; BEST-Knee Research Team. Use of Recommended Non-surgical Knee Osteoarthritis Management in Patients prior to Total Knee Arthroplasty: A Cross-sectional Study. J Rheumatol. 2020 Aug 1;47(8):1253-1260. doi: 10.3899/jrheum.190467. Epub 2019 Nov 15. PMID 31732554
- [Background] Malian, S.J., Predictors of appropriate referral to total knee arthroplasty: a validation study, in Health and Rehabilitation Sciences. 2015, Western University: Electronic Thesis and Dissertation Repository. p. 75.
- [Background] Churchill L, Malian SJ, Chesworth BM, Bryant D, MacDonald SJ, Marsh JD, Giffin JR. The development and validation of a multivariable model to predict whether patients referred for total knee replacement are suitable surgical candidates at the time of initial consultation. Can J Surg. 2016 Dec;59(6):407-414. doi: 10.1503/cjs.004316. PMID 28234616
- [Background] Pedersen BK, Saltin B. Exercise as medicine - evidence for prescribing exercise as therapy in 26 different chronic diseases. Scand J Med Sci Sports. 2015 Dec;25 Suppl 3:1-72. doi: 10.1111/sms.12581. PMID 26606383
- [Background] Lewis BS, Lynch WD. The effect of physician advice on exercise behavior. Prev Med. 1993 Jan;22(1):110-21. doi: 10.1006/pmed.1993.1008. PMID 8475007
- [Background] Andersen RE, Blair SN, Cheskin LJ, Bartlett SJ. Encouraging patients to become more physically active: the physician's role. Ann Intern Med. 1997 Sep 1;127(5):395-400. doi: 10.7326/0003-4819-127-5-199709010-00010. No abstract available. PMID 9273831
- [Background] Flores Mateo G, Granado-Font E, Ferre-Grau C, Montana-Carreras X. Mobile Phone Apps to Promote Weight Loss and Increase Physical Activity: A Systematic Review and Meta-Analysis. J Med Internet Res. 2015 Nov 10;17(11):e253. doi: 10.2196/jmir.4836. PMID 26554314
- [Background] Skou ST, Odgaard A, Rasmussen JO, Roos EM. Group education and exercise is feasible in knee and hip osteoarthritis. Dan Med J. 2012 Dec;59(12):A4554. PMID 23290290
- [Background] Skou ST, Simonsen ME, Odgaard A, Roos EM. Predictors of long-term effect from education and exercise in patients with knee and hip pain. Dan Med J. 2014 Jul;61(7):A4867. PMID 25123117
- [Background] Skou ST, Roos EM. Good Life with osteoArthritis in Denmark (GLA:D): evidence-based education and supervised neuromuscular exercise delivered by certified physiotherapists nationwide. BMC Musculoskelet Disord. 2017 Feb 7;18(1):72. doi: 10.1186/s12891-017-1439-y. PMID 28173795
- [Background] Maksymowych WP, Richardson R, Mallon C, van der Heijde D, Boonen A. Evaluation and validation of the patient acceptable symptom state (PASS) in patients with ankylosing spondylitis. Arthritis Rheum. 2007 Feb 15;57(1):133-9. doi: 10.1002/art.22469. PMID 17266072
- [Background] Agarwal P, Kithulegoda N, Bouck Z, Bosiak B, Birnbaum I, Reddeman L, Steiner L, Altman L, Mawson R, Propp R, Thornton J, Ivers N. Feasibility of an Electronic Health Tool to Promote Physical Activity in Primary Care: Pilot Cluster Randomized Controlled Trial. J Med Internet Res. 2020 Feb 14;22(2):e15424. doi: 10.2196/15424. PMID 32130122
- [Background] Keating XD, Zhou K, Liu X, Hodges M, Liu J, Guan J, Phelps A, Castro-Pinero J. Reliability and Concurrent Validity of Global Physical Activity Questionnaire (GPAQ): A Systematic Review. Int J Environ Res Public Health. 2019 Oct 26;16(21):4128. doi: 10.3390/ijerph16214128. PMID 31717742
- [Background] Dobson F, Hinman RS, Hall M, Terwee CB, Roos EM, Bennell KL. Measurement properties of performance-based measures to assess physical function in hip and knee osteoarthritis: a systematic review. Osteoarthritis Cartilage. 2012 Dec;20(12):1548-62. doi: 10.1016/j.joca.2012.08.015. Epub 2012 Aug 31. PMID 22944525
- [Background] Klassbo M, Larsson E, Mannevik E. Hip disability and osteoarthritis outcome score. An extension of the Western Ontario and McMaster Universities Osteoarthritis Index. Scand J Rheumatol. 2003;32(1):46-51. doi: 10.1080/03009740310000409. PMID 12635946
- [Background] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558
- [Background] Hawker GA, Davis AM, French MR, Cibere J, Jordan JM, March L, Suarez-Almazor M, Katz JN, Dieppe P. Development and preliminary psychometric testing of a new OA pain measure--an OARSI/OMERACT initiative. Osteoarthritis Cartilage. 2008 Apr;16(4):409-14. doi: 10.1016/j.joca.2007.12.015. PMID 18381179
- [Background] Hawker GA, Stewart L, French MR, Cibere J, Jordan JM, March L, Suarez-Almazor M, Gooberman-Hill R. Understanding the pain experience in hip and knee osteoarthritis--an OARSI/OMERACT initiative. Osteoarthritis Cartilage. 2008 Apr;16(4):415-22. doi: 10.1016/j.joca.2007.12.017. Epub 2008 Mar 4. PMID 18296075
- [Background] Scott PJ, Huskisson EC. Measurement of functional capacity with visual analogue scales. Rheumatol Rehabil. 1977 Nov;16(4):257-9. doi: 10.1093/rheumatology/16.4.257. PMID 414343
- [Background] Balestroni G, Bertolotti G. [EuroQol-5D (EQ-5D): an instrument for measuring quality of life]. Monaldi Arch Chest Dis. 2012 Sep;78(3):155-9. doi: 10.4081/monaldi.2012.121. Italian. PMID 23614330
- [Background] Lorig K, Chastain RL, Ung E, Shoor S, Holman HR. Development and evaluation of a scale to measure perceived self-efficacy in people with arthritis. Arthritis Rheum. 1989 Jan;32(1):37-44. doi: 10.1002/anr.1780320107. PMID 2912463
- [Background] Radloff, L.S., The CES-D Scale:A Self-Report Depression Scale for Research in the General Population. Applied Psychological Measurement, 1977. 1(3): p. 385-401.
- [Background] Lee KA, Hicks G, Nino-Murcia G. Validity and reliability of a scale to assess fatigue. Psychiatry Res. 1991 Mar;36(3):291-8. doi: 10.1016/0165-1781(91)90027-m. PMID 2062970
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Braun, V. and V. Clarke, Using thematic analysis in psychology. Qualitative Research in Psychology, 2006. 3(2): p. 77-101.
- [Derived] Thornton J, Barton KI, Churchill L, Schulz JM, Bryant D, Ambrose A, Hart HF, Stephenson D, Zou G, Correa S, MacDonald SJ, Degen R, Zwarenstein M, Getgood A. Novel uses of healthcare technology for individuals with mild to moderate hip or knee osteoarthritis: The technology, exercise and activity prescription for enhanced mobility (TEAM) study randomized controlled trial protocol. Osteoarthr Cartil Open. 2025 Feb 25;7(2):100586. doi: 10.1016/j.ocarto.2025.100586. eCollection 2025 Jun. PMID 40115196